| The Effectiveness of Game-Based Virtual Reality Approach in Patients with |
|---------------------------------------------------------------------------|
| Subacromial Impingement Syndrome |

Study Protocol and Statistical Analysis Plan (SAP)

(Pages 1 - 20)

| The Effectiveness of Game-Based Virtual Reality Approach in Patient | s with |
|---------------------------------------------------------------------|--------|
| Subacromial Impingement Syndrome | |

**Study Protocol** 

(Pages 2 – 5)

## **Study Protocol**

Study titled "The Effectiveness of Game-Based Virtual Reality Approach in Patients with Subacromial Impingement Syndrome" was approved by Marmara University Faculty of Health Sciences Ethical Committee at the meeting on 29.11.2018 with approval number: 36 (Annex-1).

The legal representatives of the patients who participated in the study will be informed about the aim, duration and the programs to be applied throughout the study. Volunteer Information Form will be signed and approved in accordance with the standards deemed appropriate by the Ethical Committee of Marmara University Faculty of Health Sciences. The study will be conducted in accordance with the Declaration of Helsinki.

## **Hypothesis of the Study**

H<sub>0</sub>: Addition of game-based virtual reality exercises to the rehabilitation program in patients with subacromial impingement syndrome does not contribute positively in improving the effectiveness of upper extremity for pain, range of motion and disability

H<sub>1</sub>: Addition of game-based virtual reality exercises to the rehabilitation program in patients with subacromial impingement syndrome contribute positively in improving the effectiveness of upper extremity for pain, range of motion and disability.

## Randomization of the Study Groups

Individuals with Subacromial Impingement Syndrome applying to Cadde Medical Center for treatment will be invited to participate in the study. Individuals who volunteered to participate and whom met the criteria for participation will be randomized with simple random sampling method and will be divided into two groups. In both groups participants will receive conventional physiotherapy and rehabilitation. In the study group, 10 minutes of exercises with the game-based virtual reality exercises will added to the conventional physiotherapy and rehabilitation methods

### **Inclusion Criteria**

- Volunteered to participate in the study,
- Aged between 18-65 years

### **Exclusion Criteria**

- Any visual or hearing problem,
- Other neurological, orthopedic or rheumatic problems that may restrict shoulder motion or cause pain,
- Having a physical disability or uncontrolled chronic systemic disease,
- Major trauma,
- Treatment for shoulder problems within the last 6 months,
- History of epilepsy

### **Evaluations**

A Physiotherapist will applying the following evaluation parameters at the baseline, and at the end of 4-weeks treatment program, the same physiotherapist will be applying evaluation parameters. Primary outcome measures and applied evaluations are shown in Table 1.

**Table 1.** Primary outcome measures and evaluation methods

| Primary Outcome Measures | Evaluation Methods |
|---|---|
| Range of Motion (ROM) | Goniometer |
| Pain | Visual Analogue Scale (VAS) |
| Disability | The Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire |
| Quality of Shoulder Function | Constant-Murley Score |
| Muscle Strength | Dynomometer |
| Pain Threshold | Algometer |
| Proprioception | Marmara Visual Auditory Joint Education Device (MarvaJED) |
| Kinesiophobia | Tampa Kinesiophobia Scale (TKS) |
| Satisfaction of the Treatment | Visual Analogue Scale (VAS) |

The range of motion will be defined with 'goniometer', the pain with 'Visual Analogue Scale (VAS)', the disability with 'The Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire', the quality of shoulder function with 'Constant- Murley Score', the muscle strength with 'dynomometer', the pain threshold with algometer, the proprioception with

'Marmara Visual Auditory Joint Education Device (MarvaJED)', the kinesiophobia with 'Tampa Kinesiophobia Scale (TKS), the satisfaciton of the treatment with 'Visual Analog Scale (VAS)'.

## **Treatment Program**

The participants in the study will be rehabilitated in Cadde Medical Center for 5 times a week for 4 weeks, a total of 20 sessions (Duration of one session is 60 minutes).

Group I (Control Group) will receive conventional physiotherapy and rehabilitation treatment program

Group II (Study Group) will receive conventional physiotherapy and rehabilitation treatment program and game-based virtual reality exercises (with a device named USE-IT) (10 minutes).

## **Game-Based Virtual Reality Exercises**

In addition to the conventional physiotherapy and rehabilitation program, a 10-minute game-based virtual reality exercises will be applied. A game-based virtual reality device named USE-IT will be added to the rehabilitation program. USE-IT is a technological rehabilitation system designed by the Department of Physiotherapy and Rehabilitation at Hacettepe University (Ankara, Turkey). It is a smart gaming device which has been used in patients who suffer from movement loss in their upper extremities due to various neurological and orthopedic reasons.

## **Conventional Physiotherapy and Rehabilitation Program**

The conventional physiotherapy and rehabilitation program includes the application of Transcutaneous Electrical Nerve Stimulation (TENS), cold pack, therapeutic ultrasound, Codman Exercises, Wand exercises, shoulder wheel exercises, finger ladder exercises, strengthening exercises with elastic band and capsule stretching.

| The Effectiveness of Game-Based Virtual Reality Approach in Patients w | vith |
|---|---|
| Subacromial Impingement Syndrome | |

Statistical Analysis Plan (SAP)

(Pages 6 – 7)

## **Statistical Analysis Plan (SAP)**

The statistical program Statistical Package for Social Sciences (SPSS) Version 11.5 (SPSS Inc., Chicago, IL, USA) will be used in the data analysis of the study. The p value of p<0.05 will be considered to be statistically significant in the data analysis. The initial demographic characteristics (age, boy, body weight) of all patients included in the study will be calculated.

'Shaphiro-Wilks Test' will be used to investigate the appropriateness of the variables to normal distribution. 't-test' will be used to compare the parameters of normal distribution in order to investigate the efficacy studies before and after the treatment; 'Wilcoxon Test' will be used to compare the parameters that do not comply with normal distribution.

| The Effectiveness of Game-Based Virtual Reality Approach in Patients w | vith |
|---|---|
| Subacromial Impingement Syndrome | |

Annex

(Pages 8 – 20)

# Annex 1. Marmara University Faculty of Health Sciences Ethical Committee Approval (Approval made at the meeting on 29.11.2018 with number: 36)



# MARMARA ÜNİVERSİTESİ Sağlık Bilimleri Fakültesi Girişimsel Olmayan Etik Kurulu

PROJENÍN ADI

ROJENÍN YŪRŪTÜCÜSÜ PROJEDEKİ ARAŞTIRICILAR ONAY TARİHİ VE SAYISI

: "Subakromiyal Sıkışma Sendromlu Olgularda Oyun Temelli

Sanal Gerçeklik Yaklaşımının Etkinliği"

: Doç. Dr. Zübeyir SARI

: Berivan Beril KILIÇ, Dilara Merve SARI, Nimet SERMENLİ

Prof. Dr. M. G Etik Kurul Baş

: 29.11.2018/36

Sayın: Doç. Dr. Zübeyir SARI

"36" protokol numaralı "Subakromiyal Sıkışma Sendromlu Olgularda Oyun Temelli Sanal Gerçeklik Yaklaşımının Etkinliği" isimli projeniz Fakültemiz Etik Kurulu tarafından incelenmiş oy birliği ile etik yönden uygun olduğuna karar verilmiştir.

Prof. Dr. Mehy

Prof. Dr. Ayşen GARGILI

Dog Dr. M. Barrin BLSAHIN

Doç. Dr. Ş. Burak BEKAROĞLU

Doç. Dr. Zübeyir SARI

r. MeltemBAL

Doc. Dr. Saime EROL

Dr. Öğr. Üyesi Murat D.

Dr. Öğr. Üyesi K. Burcu ÇALIK

Dr. Öğr. Üyesi Ayşe KARAKQÇ

Dr. Öğr. Üyesi Şule

AKTAÇ

Dr. Öğr. Üyesi S. Kumral ÖZÇELİK









# Annex 2. Participants Tracking Form

| Name-Surn | name: | | Date: |
|---|---|---|---|
| Tel Numbe | r: | | Birth Date: |
| Age: | Sex: | Height: | Weight: |
| Dominant S | Side (Mark): Rig | ht / Left | |
| Effected Si | de (Mark): Rig | ght/ Left | |
| How did th | e problem occur | ? (Please explain): | |
| Did you ha | ve any operation | ? Please write, if you | did: |
| Do you hav | e any additional | problem? | |
| No: | | | |
| Yes/ If yes, | What is it? | | |
| | Asses | sment of Pain - Visua | l Analogue Scale |
| - How | v severe is your sh | oulder pain during acti | vity? |
| | | 5 | |
| (no pain) | | | (worst possible pain) |
| - How | severe is your sh | oulder pain during rest | ? |
| | | 5 | |
| (no pain) | | | (worst possible pain) |

# Assessment of Range of Motion and Muscle Strength

| | Muscle Strength | | | Range of Motion | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | R | | L | | | R | | L | | |
| | 1 | 2 | 1 | 2 | 1 | 2 | 3 | 1 | 2 | 3 |
| Shoulder | | | | | | | | | | |
| Flexion | | | | | | | | | | |
| Shoulder | | | | | | | | | | |
| Extension | | | | | | | | | | |
| Shoulder | | | | | | | | | | |
| Abduction | | | | | | | | | | |
| Shoulder | | | | | | | | | | |
| Adduction | | | | | | | | | | |
| Shoulder<br>IR | | | | | | | | | | |
| Shoulder<br>ER | | | | | | | | | | |
| Elbow<br>Flexion | | | | | | | | | | |
| Elbow<br>Extension | | | | | | | | | | |
| Supination | | | | | | | | | | |
| Pronation | | | | | | | | | | |

# Assesment of Disability - Disabilities of the Arm, Shoulder and Hand Questionnaire—DASH

# DISABILITIES OF THE ARM, SHOULDER AND HAND - British English

Please rate your ability to do the following activities in the last week by circling the number below the appropriate response.

| | NO | MILD | MODERATE | SEVERE | UNABLE |
|---|---|---|---|---|---|
| | DIFFICULTY | DIFFICULTY | DIFFICULTY | DIFFICULTY | |
| 1 Open a tight or new jar | 1 | 2 | 3 | 4 | 5 |
| 2 Write | 1 | 2 | 3 | 4 | 5 |
| 3 Turn a key | 1 | 2 | 3 | 4 | 5 |
| 4 Prepare a meal. | 1 | 2 | 3 | 4 | 5 |
| 5 Push open a heavy door | 1 | 2 | 3 | 4 | 5 |
| 6 Place an object on a shelf above your head | 1 | 2 | 3 | 4 | 5 |
| 7 Do heavy household jobs (e.g. wash windows, clean floors) | 1 | 2 | 3 | 4 | 5 |
| 8 Garden or outdoor property work | 1 | 2 | 3 | 4 | 5 |
| 9 Make a bed | 1 | 2 | 3 | 4 | 5 |
| 10 Cary a shopping bag or briefcase | 1 | 2 | 3 | 4 | 5 |
| 11 Carry a heavy object (over 10 lbs/ 5kgs) | 1 | 2 | 3 | 4 | 5 |
| 12 Change a lightbulb overhead | 1 | 2 | 3 | 4 | 5 |
| 13 Wash or blow dry your hair | 1 | 2 | 3 | 4 | 5 |
| 14 Wash your back | 1 | 2 | 3 | 4 | 5 |
| 15 Put on a jumper | 1 | 2 | 3 | 4 | 5 |
| 16 Use a knife to cut food | 1 | 2 | 3 | 4 | 5 |
| 17 Recreational activities which require little effort (e.g. card playing, knitting, etc) | 1 | 2 | 3 | 4 | 5 |
| 17 Recreational activities which require you to take some force or impact through your arm, shoulder or hand (e.g. golf, hammering, tennis etc) | 1 | 2 | 3 | 4 | 5 |
| 18 Recreational activities in which you move your arm freely (e.g. playing Frisbee, badminton etc) | 1 | 2 | 3 | 4 | 5 |
| 20 Manage transport needs (getting from one place to another) | 1 | 2 | 3 | 4 | 5 |
| 21 Sexual activities | 1 | 2 | 3 | 4 | 5 |

| | NOT AT<br>ALL | SUGHTLY | MODERATELY | Quite a<br>bit | Extremely |
|---|---|---|---|---|---|
| 22 During the past week, to what extent has your arm, shoulder or hand problem interfered with your normal social activities with family. friends, neighbours or groups? (circle number) | 1 | 2 | 3 | 4 | 5 |
| | NOT<br>LIMITED AT<br>ALL | SUGHTLY | MODERATELY<br>LIMITED | VERY<br>LIMITED | UNABLE |
| 23 During the past week, were you limited in your work or other regular daily activities as a result of your arm, shoulder or hand problem? (circle number) | 1 | 2 | 3 | 4 | 5 |
| Please rate the severity of the following symptoms in the last week (circle number) | NONE | MILD | MODERATE | SEVERE | EXTREME |
| 24 Arm, shoulder or hand pain | 1 | 2 | 3 | 4 | 5 |
| 25 Arm, shoulder or hand pain when you do any specific activity | 1 | 2 | 3 | 4 | 5 |
| 26 Tingling (pins and needles) in your arm, shoulder or hand | 1 | 2 | 3 | 4 | 5 |
| 27. Weakness in your arm, shoulder or hand | 1 | 2 | 3 | 4 | 5 |
| 28 Stiffness in your arm, shoulder or hand | 1 | 2 | 3 | 4 | 5 |
| | NO<br>DIFFICULTY | MILD<br>DIFFICULT<br>Y | MODERATE<br>DIFFCULTY | SEVERE<br>DIFFCULT<br>Y | SO MUCH DIFFICULTY THAT I CAN'T SLEEP |
| 29 During the past week, how much difficulty have you had sleeping because of the pain in your arm, shoulder or hand? (circle number) | 1 | 2 | 3 | 4 | 5 |
| | STRONGLY<br>DISAGREE | DISAGREE | NEITHER AGREE<br>OR DISAGREE | AGREE | STRONGLY<br>AGREE |
| 30 I feel less capable, less confident or less useful because of my arm, shoulder or hand problem (circle number) | 1 | 2 | 3 | 4 | 5 |

DASH DISABILITY/SYMPTOM SCORE = [(sum of n responses)-1] x 25 (where n is the number of completed responses)

A DASH score may not be calculated if there are greater than 3 missing items.

3

# DISABILITIES OF THE ARM, SHOULDER AND HAND - British English

#### WORK MODULE (OPTIONAL)

The following questions ask about the impact of your arm, shoulder or hand problem on your ability to work (including home-making if that is your main work role).

Please indicate what your job / work is:

☐ I do not work (you may skip this section).

Please circle the number that best describes your physical ability in the past week. Did you have any difficulty:

| | | NO<br>DIFFICULTY | MILD<br>DIFFICULTY | MODERATE<br>DIFFICULTY | SEVERE<br>DIFFICULTY | UNABLE |
|---|---|---|---|---|---|---|
| 1. | Doing your work in your usual way? | 1 | 2 | 3 | 4 | 5 |
| 2. | Doing your usual work because of arm, shoulder or hand pain? | 1 | 2 | 3 | 4 | 5 |
| 3. | Doing your work as well as you would like? | 1 | 2 | 3 | 4 | 5 |
| 4. | Spending your usual amount of time doing your work? | 1 | 2 | 3 | 4 | 5 |

### SPORTS/PERFORMING ARTS MODULE (OPTIONAL)

The following questions relate to the impact of your arm, shoulder or hand problem on playing *your musical instrument or sport or both*. If you play more than one sport or instrument (or play both), please answer with respect to that activity which is most important to you.

Please indicate the sport or instrument which is most important to you: \_\_\_\_\_\_\_

☐ I do not play a sport or an instrument. (You may skip this section).

Please circle the number that best describes your physical ability in the past week. Did you have any difficulty:

| | | NO<br>DIFFICULTY | MILD<br>DIFFICULTY | MODERATE<br>DIFFICULTY | SEVERE<br>DIFFICULTY | UNABLE |
|---|---|---|---|---|---|---|
| 1. | Playing your instrument or sport in your usual way? | 1 | 2 | 3 | 4 | 5 |
| 2. | Playing your musical instrument or sport because of arm, shoulder or hand pain? | 1 | 2 | 3 | 4 | 5 |
| 3. | Playing your instrument or sport as well as you would like? | 1 | 2 | 3 | 4 | 5 |
| 4. | Spending your usual amount of time<br>practising or playing your instrument or<br>sport? | 1 | 2 | 3 | 4 | 5 |

Scoring the optional modules: add up the assigned values for each response;

Divide by 4 (number of items); subtract 1; multiple by 25.

An optional module score may <u>not</u> be calculated if there are any missing items.

4

# **Assessment of Quality of Shoulder Function- Constant Murley Score**

# Patient-based Questionnaire

| | Date: |
|---|---|
| PATI | IENT'S NAME: PATIENT NUMBER: |
| We v | would be grateful if you could take a few minutes to fill in this questionnaire. It is an essential part of our uation of the results of our treatment and surgery. It ultimately improves the quality of service we provide to PLEASE COMPLETE THE FORM BY CIRCLING THE MOST APPROPRIATE RESPONSE. |
| Α. | PAIN A1. Do you have pain in your shoulder during normal activities? (Please circle the most appropriate response) |
| | 1. NO PAIN 2. MILD PAIN 3. MODERATE PAIN 4. SEVERE PAIN |
| 0 | A2. LEVEL OF PAIN If 0 means no pain and 15 means the worst pain you can have, please circle the number which describes your shoulder pain when you are doing normal activities: 0 1 2 3 4 5 6 7 8 9 10 11 12 13 14 15 ® NONE MILD MODERATE SEVERE UNBEARABLE |
| В. | B1. Does your shoulder limit your occupation or daily living? 1. NO OR VERY SLIGHTLY 2. MODERATE LIMITATION B2. Are your leisure and recreational activities limited by your shoulder? 1. NO OR VERY SLIGHTLY 2. MODERATE LIMITATION 3. SEVERE LIMITATION |
| | B3. Does your shoulder disturb your night sleep? 1. NO 2. SOMETIMES 3. YES |
| | B4. What level can you use your arm for reasonable painless movement? |
| | 1. WAIST 2. CHEST 3. NECK 4. EAR 5. ABOVE HEAD |

B5. On a scale of 0 to 10, where **0** is **not satisfied** and **10** is **very satisfied**, how satisfied are you with your shoulder? **(Circle the correct number)** 

80 1 2 3 4 5 6 7 8 9 10

| C. <u>vv</u> | HAT IS TOOK OCCUPA | 110N F | | |
|---|---|---|---|---|
| | C1. How well can you | perform your occup | ation? (Pleas | e circle the most appropriate response) |
| | 1. EASILY | 2. WITH LITTLE D | IFFICULTY | 3. WITH MODERATE DIFFICULTY |
| | 4. WITH EXTRE | ME DIFFICULTY | 5. N | OT AT ALL |
| | C2. What are your tw | o main sporting/leis | ure activities | , |
| | C3. How well can you | perform these activ | ities? (Please | circle the most appropriate response) |
| | 1. EASILY | 2. WITH LITTLE D | DIFFICULTY | 3. WITH MODERATE DIFFICULTY |
| | 4. WITH EXTRE | ME DIFFICULTY | 5. NOT A | T ALL |
| ==== | | | | if you have had an operation |
| D. FC | | | | |
| | | | | ration:] |
| | D1. How do you feel in (Please circle the | now, following your o<br>most appropriate re | • | |
| | 1. MUCH BETTER | 2. BETTER | 3. SAME | 4. WORSE |
| | | Please circle the mos | | e response) |
| | 2. Returned to the same occupation but with decreased level of activity (due to the shoulder) | | | |
| | 3. Changed occupation due to the shoulder? | | | |
| | 4. Stopped working altogether because of your shoulder? | | | |
| | D3. If you have chang | ed occupation, what | | o now?: |
| | D4. Have you now (PI | ease circle the most | appropriate | response) |
| | 1. Returned to | the same level of act | tivity in the sa | ame sport? |
| | 2. Returned to | a decreased level of | activity in the | e same sport (because of the shoulder)? |
| | 3. Changed spo | orts because of the sl | houlder? | |
| | 4. Stopped plan | ying sports altogethe | | |
| | , | , | , | |

## E. Range of Motion

Copy the movements the model is performing – it may be useful to perform this exercise in front of a mirror.

Starting from left to right in each row

- Tick the box (below each photograph) if you are able to perform the action
- . Leave the box blank if you cannot perform the action



### F. Strength

Look at the two photographs below. Try to hold your arm in this position for 3 seconds each time carrying weights in the plastic bag.

Please use as weights within the plastic bag:

- Bags of sugar
- and/or
- · Filled plastic bottles of milk (may be filled with water)

and/or

· Whatever is available for you with known weight

Please record in the spaces below what was the maximum weight in kilograms (or pounds) or litres (or pints) that you were able to hold in this position for 3 seconds for each arm.



Seen from the front



seen from above

The maximum weight that I was able to hold in this position for 3 seconds:

| Right Arm: | Kilograms/Litres | Left Arm: | Kilograms/Litres |
|------------|------------------|-----------|------------------|
| Right Arm: | Pounds/Pints | Left Arm: | Pounds/Pints |

## G. COMMENTS

The space below is for any further comments you would like to make.

Thank you for filling in this questionnaire.

# Assessment of Kinesiophobia - Tampa Kinesiophobia Scale (TKS)

# Tampa Scale for Kinesiophobia (Miller, Kori and Todd 1991)

- 1 = strongly disagree
- 2 = disagree
- 3 = agree
- 4 = strongly agree

| 1. I'm afraid that I might injury myself if I exercise | 1 | 2 | 3 | 4 |
|---|---|---|---|---|
| If I were to try to overcome it, my pain would | 1 | 2 | 3 | 4 |
| | 1 | | 3 | 4 |
| increase | | _ | 2 | |
| My body is telling me I have something | 1 | 2 | 3 | 4 |
| dangerously wrong | | | | |
| <ol> <li>My pain would probably be relieved if I were to</li> </ol> | 1 | 2 | 3 | 4 |
| exercise | | | | |
| <ol><li>People aren't taking my medical condition</li></ol> | 1 | 2 | 3 | 4 |
| seriously enough | | | | |
| 6. My accident has put my body at risk for the rest | 1 | 2 | 3 | 4 |
| of my life | | | | |
| 7. Pain always means I have injured my body | 1 | 2 | 3 | 4 |
| Just because something aggravates my pain does | 1 | 2 | 3 | 4 |
| not mean it is dangerous | _ | _ | | . |
| I am afraid that I might injure myself | 1 | 2 | 3 | 4 |
| accidentally | 1 | | 3 | 4 |
| 10. Simply being careful that I do not make any | 1 | 2 | 3 | 4 |
| | 1 | | 3 | 4 |
| unnecessary movements is the safest thing I can | | | | |
| do to prevent my pain from worsening | _ | | _ | |
| 11. I wouldn't have this much pain if there weren't | 1 | 2 | 3 | 4 |
| something potentially dangerous going on in my | | | | |
| body | | | | |
| 12. Although my condition is painful, I would be | 1 | 2 | 3 | 4 |
| better off if I were physically active | | | | |
| <ol><li>Pain lets me know when to stop exercising so</li></ol> | 1 | 2 | 3 | 4 |
| that I don't injure myself | | | | |
| 14. It's really not safe for a person with a condition | 1 | 2 | 3 | 4 |
| like mine to be physically active | | | | |
| 15. I can't do all the things normal people do | 1 | 2 | 3 | 4 |
| because it's too easy for me to get injured | * | _ | | • |
| 16. Even though something is causing me a lot of | 1 | 2 | 3 | 4 |
| pain, I don't think it's actually dangerous | 1 | | 3 | 4 |
| | 1 | _ | 2 | |
| 17. No one should have to exercise when he/she is in | 1 | 2 | 3 | 4 |
| pain | | | | |

# Assessment of satisfaction after the treatment

| - How satisfied are you with the decreas | se of pain at the end of treatment |
|---|---|
| 05 | 10 |
| (Not satisfied at all) | (Very satisfied) |
| - How satisfied are you with your functi | onality at the end of treatment? |
| 05 | 10 |
| (Not satisfied at all) | (Very satisfied) |
| - How satisfied are you with all of your | treatment? |
| 05 (Not satisfied at all) | 10 (Very satisfied) |
| - How satisfied are you with your physic | otherapist? |
| 05 | 10 |
| (Not satisfied at all) | (Very satisfied) |